CLINICAL TRIAL: NCT02359591
Title: The Development of Child Development Checklist Multimedia System and Its Clinical Evaluation
Status: Completed | Type: Observational
Sponsor: Hsin-Yi Kathy Cheng (Other)
Responsible Party: Sponsor-Investigator, Hsin-Yi Kathy Cheng, associate professor, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Other Study IDs: ChangGungMH
Record Dates: First submitted 2014-11-05; First posted 2015-02-10 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Child Development Checklist
MeSH Terms: interventions — Multimedia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- text-based or multimedia: Subject fills in a questionnaire regarding whether the child meets developmental milestones for his/her developmental age, both the text-based and the multimedia version. A total score will be calculated and compared.
  Interventions: Other: text-based or multimedia

INTERVENTIONS:
Other: text-based or multimedia — subjects fills in a questionnaire regarding whether the child meets the developmental milestones for his/her developmental age.

SUMMARY:
【Background& Purpose】In order to early detect the problems a child might have during his/her development, an effective screening tool is of great needs. The [Taipei City Child Development Screening checklist] is often used to serve this process. This text version is mainly distributed to the parents to fill out during their child regular check-ups to the hospitals and clinics. The drawbacks of this checklist is that it lacks of active participation of the target population, and the text version limits its usage to people who are not familiar with Chinese characteristics, such as those new inhabitant. These lead to low screening rates therefore causing delayed early intervention. 【Purpose】The purpose of this study was to design and develop the multi-media graphic version of the [Taipei City Child Development Screening checklist] based on its original text version.【Method】The developed muti-media system will be checked for is validity. Thirty parents/legal guardians of children in each target age groups will be recruited randomly for the clinical reliability evaluation.

ELIGIBILITY:
Inclusion Criteria:

* For parents/primary caregivers whose children are between 3 months and 7 years old can participate.

Exclusion Criteria:

* Any visual impairment.

Ages: 20 Months to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: guardians whose child is between 3 months and 7 years old
Sampling Method: Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2014-03; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
13 developmental milestones questionnaire | baseline
  there will be 13 developmental milestones in each age range. The guardian of each subject check "yes/no" depends on whether his/her child reaches the milestone

CONTACTS AND LOCATIONS:
Overall Officials: Chang Gung Medical Hospital Chang Gung Medical Hospital, Study Director — Chang Gung Medical Hospital
Locations (1):
- Chang Gung Univ., Taoyuan District, Taiwan

REFERENCES:
- [Derived] Cheng HK, Chen LY, Cheng CH, Ju YY, Chen CL, Tseng KC. A Multimedia Child Developmental Screening Checklist: Design and Validation. J Med Internet Res. 2016 Oct 24;18(10):e277. doi: 10.2196/jmir.6249. PMID 27777218